CLINICAL TRIAL: NCT01709409
Title: A Randomized, Controlled, Partially Double-blinded, Phase 3, Multi-center Trial to Determine if Curosurf® Reduces the Duration of Mechanical Ventilation in Infants 24+0 to 31+6 Weeks Gestational Age
Brief Title: A Multi-center Trial to Determine if Curosurf® Reduces the Duration of Mechanical Ventilation in Very Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Curosurf-01
Record Dates: First submitted 2012-10-12; First posted 2012-10-18 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-06

CONDITIONS: Respiratory Distress Syndrome
Keywords: Prematurity
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Curosurf (Group 1) (Experimental): Surfactant(Curosurf in this arm) is given for treatment of RDS after the diagnosis has been made by the Neonatologist. The treatment dose for Curosurf® is 2.5 ml/kg (200mg/kg) for the first dose and 1.25 ml/kg (100mg/kg) for repeat doses, given by endotracheal method. There is a maximum of 3 doses in the study.
  Interventions: Drug: Curosurf-Group1
- BLES (Group 2) (Active Comparator): Surfactant(BLES in this arm) is given for treatment of RDS after the diagnosis has been made by the Neonatologist. For BLES the recommended dose is 5 ml/kg. given by endotracheal method. There is a maximum of 3 doses in the study.
  Interventions: Drug: BLES-group 2

INTERVENTIONS:
Drug: Curosurf-Group1 — Maximum of 3 doses are administered to infants diagnosed with RDS.
  Arms: Curosurf (Group 1)
Drug: BLES-group 2 — Maximum of 3 doses are administered to infants with RDS
  Arms: BLES (Group 2)

SUMMARY:
The purpose of this study is to see if a medication called Curosurf can reduce the length of time that small premature babies with Respiratory Distress Syndrome (immature lungs) or RDS, stay on the ventilator, as compared to the standard medication called BLES. Curosurf is a medication that is already used in other countries around the world but not yet in Canada.

Babies born under 32 weeks of gestation frequently need respiratory support after birth, including being placed on a breathing machine or respirator. The most common reason is Respiratory Distress Syndrome (RDS) whereby immature lungs don't produce enough surfactant, a soapy like substance that helps the air sacs open and close. Our current standard treatment is a surfactant called BLES. Curosurf contains more active ingredient per volume therefore the amount is smaller. The investigators hypothesize that babies who receive Curosurf will be able to be removed from the ventilator sooner.

Babies in this study will have a 50/50 chance of receiving either Curosurf or BLES and the investigators will monitor their progress during their Neonatal Intensive Care Unit admission.

The study is taking place in Canada. The goal is to enroll 88 babies. There are no extra tests (blood tests or X-Rays) or return visits to the hospital for the purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born between 24+0 and 31+6 weeks gestational age, admitted to the study centers
2. Infants with RDS requiring intubation and surfactant therapy within 48 hours after birth

Exclusion Criteria:

1. Any infant more than 48 hours of age
2. Any infant with a pulmonary hemorrhage
3. Any infant with life-threatening congenital anomaly or one that is considered non-viable
4. Any infant on rescue high frequency ventilation
5. Any infant known to require early intubation and ventilation for surgical treatment of a congenital anomaly
6. Any infant with anomalies of the upper or lower airway or mandible precluding use of nCPAP
7. Any infant born after prolonged premature rupture of membranes (<22 weeks GA or >28 days prior to delivery)
8. A parent/LAR who is incapable of, or unwilling, to give consent
9. Participation in another clinical trial of any placebo, drug, biological, or device conducted under the provisions of a protocol
10. Any other reason as deemed significant by the Investigator

Ages: 24 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2013-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Lemyre, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lemyre B, Fusch C, Schmolzer GM, Rouvinez Bouali N, Reddy D, Barrowman N, Huneault-Purney N, Lacaze-Masmonteil T. Poractant alfa versus bovine lipid extract surfactant for infants 24+0 to 31+6 weeks gestational age: A randomized controlled trial. PLoS One. 2017 May 4;12(5):e0175922. doi: 10.1371/journal.pone.0175922. eCollection 2017. PMID 28472058
- See also: Product information — http://www.curosurf.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three university-affiliated tertiary NICUs recruited patients between March 2013 and December 2015. 560 patients were screening for eligibility.
Pre-assignment Details: One patient in the Curosurf group was found to have an exclusion criteria after randomization and was excluded (he did not receive the assigned treatment).
Groups:
- Curosurf (Group 1): Surfactant(Curosurf in this arm) was given for treatment of established RDS. The treatment dose for Curosurf® was 2.5 ml/kg (200mg/kg) for the first dose and 1.25 ml/kg (100mg/kg) for repeat doses, given by endotracheal method. There was a maximum of 3 doses in the study.
- BLES (Group 2): Surfactant(BLES in this arm) was given for treatment of established RDS. The treatment dose for BLES was 5 ml/kg. given by endotracheal method. There was a maximum of 3 doses in the study.
Period: Overall Study
Arm/Group | Curosurf (Group 1) | BLES (Group 2)
Started | 43 | 45
Completed | 42 | 45
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: 1. Infants born between 24+0 and 31+6 weeks gestational age, admitted to the study centers
  2. Infants with RDS requiring intubation and surfactant therapy within 48 hours after birth
Groups:
- Total: Total of all reporting groups
Arm/Group | Curosurf (Group 1) | BLES (Group 2) | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Continuous [Mean (Standard Deviation); unit: weeks gestational age] | 26.5 (1.5) | 26.9 (2.1) | 26.7 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 35
  Male | 19 | 33 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 42 | 45 | 87
fraction of inspired oxygen [Median (Inter-Quartile Range); unit: % of inspired oxygen] | 45 [32 to 65] | 45 [35 to 50] | 45 [35 to 60]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of the Study is to Compare Between the Two Groups, the Number of Subjects Alive and Extubated at 48 Hours Post Surfactant Administration. Extubation
Description: 1. rate on ventilator ≤40 per minute and
  2. mean airway pressure ≤ 10 cm H20 and
  3. fi02 ≤ 30%
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Curosurf (Group 1) | BLES (Group 2)
Number analyzed (Participants) | 42 | 45
Participants | 21 | 26

2. Secondary Outcome: To Compare the Duration of Respiratory Support, Extubation Failure Rates, Need for Additional Surfactant Doses, Adverse Events (During and Following Administration), Survival and Pulmonary Morbidities During Hospital Admission Between the Two Groups.
Description: 1. Extubation failure
Time Frame: 36 weeks GA
Reporting Status: Not Posted

3. Secondary Outcome: Curosurf-01
Description: 2. Duration of first intubation (in hours/days)
Time Frame: 36 weeks GA
Reporting Status: Not Posted

4. Secondary Outcome: Curosurf-01
Description: 3. Total duration of respiratory support (ventilator and nCPAP) and total number of days of oxygen requirement
Time Frame: 36 weeks GA
Reporting Status: Not Posted

5. Secondary Outcome: Curosurf-01
Description: 4. Number of doses of surfactant received
Time Frame: 36 weeks GA
Reporting Status: Not Posted

6. Secondary Outcome: Curosurf-01
Description: 5. Adverse events during or after administration of surfactant
Time Frame: 36 weeks GA
Reporting Status: Not Posted

7. Secondary Outcome: Curosurf-01
Description: 6. Bronchopulmonary dysplasia, defined as oxygen or respiratory support requirement at 36 weeks corrected GA
Time Frame: 36 Weeks GA
Reporting Status: Not Posted

8. Secondary Outcome: Curosurf-01
Description: 7. Mortality prior to discharge
Time Frame: 36 weeks GA
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Curosurf (Group 1) | BLES (Group 2)
Serious Adverse Events (participants affected / at risk) | 5/42 | 11/45
Other Adverse Events (participants affected / at risk) | 1/42 | 1/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Curosurf (Group 1) (N=42) | BLES (Group 2) (N=45)
severe airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
air leak (Reproductive system and breast disorders) | 3 (3) | 5 (5)
pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
needing CPR (Cardiac disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Curosurf (Group 1) (N=42) | BLES (Group 2) (N=45)
pulmonary interstitial emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No